CLINICAL TRIAL: NCT05593510
Title: Identifying Food Pantry Client and Staff Preferences for Nutritious no Prep Ready-to-eat Meals Versus Ingredient Bundles as an Effort to Increase Food Security, Improve Nutrition, and Promote Well-being
Brief Title: Food Pantry Client and Staff Preferences for Nutritious no Prep Ready-to-eat Meals
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Texas Southwestern Medical Center (Other)
Responsible Party: Principal Investigator, Kelseanna Hollis-Hansen, Assistant Professor, University of Texas Southwestern Medical Center
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Prevention
Other Study IDs: STU-2022-0809
Record Dates: First submitted 2022-10-20; First posted 2022-10-25 (Actual); Results first posted 2025-03-11 (Actual); Last update posted 2025-03-11 (Actual); Status verified 2025-03

CONDITIONS: Diet, Healthy; Food Security
Keywords: Food security; Food pantry; Diet quality; Intervention

STUDY DESIGN:
Intervention Model Description: Randomized repeated measures between-subjects design
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- No prep ready-to-eat meals (Experimental)
  Interventions: Behavioral: No prep ready-to-eat meals
- Ingredient bundles (e.g. meal kits) (Active Comparator)
  Interventions: Behavioral: Ingredient bundles (e.g. meal kits)
- Pantry Staff Group (No Intervention): They participate in qualitative interviews only. No demographic or other identifiable information from them. They do not receive an intervention. No Intervention Group.

INTERVENTIONS:
Behavioral: No prep ready-to-eat meals — Pantry clients will select no prep ready-to-eat meals for up to 14-days' worth of meals for themselves and 2-members of their household using an online food selection platform. The food retailer supplying the meals produces over 70 meals. We have elected to study 14-days of meals to offer clients variety and determine which flavors are most desirable to clients. After ordering, meals will be retrieved from a refrigeration unit, boxed by pantry staff, and brought to the participant to take home. An example dinner is "Teriyaki Chicken with Roasted Potatoes and Broccoli", and an example breakfast is "Omelet with Peppers and Zucchini". Meals can be stored in a refrigerator or freezer and eaten immediately or after reheating depending on the meal and consumer preference.
  Arms: No prep ready-to-eat meals
Behavioral: Ingredient bundles (e.g. meal kits) — Ingredient bundles will group individual meal ingredients (e.g., chicken, teriyaki, broccoli, potatoes) in a bag or box and pair those healthy food items with a recipe that instructs the client on how to make a healthier meal. Similar to the no prep ready-to-eat meal initiative, clients will select ingredient bundles for themselves and 2-members of their household using the food pantry online food selection platform. The ingredient bundles will closely replicate the no prep ready-to-eat meals.
  Arms: Ingredient bundles (e.g. meal kits)

SUMMARY:
The specific aims of this pilot study are: Aim 1) To identify whether no prep ready to eat meals (intervention) or ingredient bundles (control) have higher client acceptability, liking, satisfaction, and perceived diet quality ratings. Aim 2) To identify whether no prep ready to eat meals (intervention) or ingredient bundles (control) have higher feasibility ratings with food pantry staff. Exploratory Aim) To identify whether no prep ready to meals (intervention) or ingredient bundles (control) lead to greater improvements in food security, perceived diet quality, and fruit and vegetable consumption.

DETAILED DESCRIPTION:
To test the first hypothesis, we will use a randomized repeated measures between-subjects design with half of the participants randomized to receive 14-days of no prep ready-to-eat meals (intervention, n=35) and half of the participants randomized to receive 14-days of ingredient bundles (control, n=35). To test the second hypothesis, we will use a mixed-methods approach with food pantry staff (N=15), including questionnaires with fixed and open-ended items on feasibility and satisfaction of each distribution strategy followed by 30-minute semi-structured 1-1 interviews conducted by UT Southwestern study staff.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older;
* ability to read, write, and speak English or Spanish;
* ability to provide informed consent;
* current or new pantry user at our community partner;
* willing to participate;
* no dietary restrictions, allergies, or sensitivities that would put the participant at-risk of harm from consuming study foods.

Exclusion Criteria:

* Under 18 years of age;
* inability to read, write, and speak English or Spanish;
* unable to provide informed consent;
* not a pantry user at our community partner or uninterested in becoming a pantry user;
* not wanting to participate;
* dietary restrictions, allergies, or sensitivities that would put the participant at-risk of harm from consuming study foods.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 85 (Actual)
Dates: Start 2023-02-12 (Actual); Primary Completion 2023-04-26 (Actual); Study Completion 2023-04-26 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Crossroads Community Services, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: Yes
We will publish the study protocol in a journal willing to publish pilot study protocols. Deidentified data will be uploaded as supplemental files along with manuscript submissions to PubMed.
Supporting Information: Study Protocol, SAP
Time Frame: Deidentified data will be available in January 2024 and will be submitted as supplemental files along with manuscript submissions to PubMed, meaning the data will be available so long as PubMed hosts supplementary data files.

REFERENCES:
- [Result] Hollis-Hansen K, Haskins C, Turcios J, Bowen ME, Leonard T, Lee M, Albin J, Wadkins-Chambers B, Thompson C, Hall T, Pruitt SL. A pilot randomized controlled trial comparing nutritious meal kits and no-prep meals to improve food security and diet quality among food pantry clients. BMC Public Health. 2023 Dec 1;23(1):2389. doi: 10.1186/s12889-023-17355-3. PMID 38041070
- [Derived] Hollis-Hansen K, Haskins C, Turcios J, Bowen ME, Leonard T, Lee M, Albin J, Chambers BW, Thompson C, Hall T, Pruitt SL. A pilot randomized controlled trial comparing nutritious meal kits and no-prep meals to improve food security and diet quality among food pantry clients. Res Sq [Preprint]. 2023 Oct 6:rs.3.rs-3029813. doi: 10.21203/rs.3.rs-3029813/v1. PMID 37886450

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Out of the total 85 participants enrolled, 70 were pantry clients that are part of the RCT, 15 pantry staff were not part of this RCT. Pantry staff group (No intervention Group) participated in qualitative interviews (anonymous) only. No demographic or other identifiable information were collected from them. They were not randomized. They did not receive an intervention.
Groups:
- Pantry Staff Group: Pantry staff only completed anonymous interviews during the study pilot. They participated in qualitative interviews only. They were not randomized. They did not receive an intervention.
Period: Overall Study
Arm/Group | No Prep Ready-to-eat Meals | Ingredient Bundles (e.g. Meal Kits) | Pantry Staff Group
Started | 35 | 35 | 15
Completed | 31 | 35 | 15
Not Completed | 4 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Pantry staff Group (15 count) is not included in Baseline Characteristics since any demographic or other identifiable information were not collected from them. They completed anonymous interviews only. They were not randomized. They did not receive an intervention.
Groups:
- Total: Total of all reporting groups
Arm/Group | No Prep Ready-to-eat Meals | Ingredient Bundles (e.g. Meal Kits) | Total
Number analyzed (Participants) | 35 | 35 | 70
Age, Continuous [Mean (Standard Deviation); unit: years] | 56.71 (13.48) | 60.43 (13.71) | 58.57 (13.62)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 31 | 32 | 63
  Male | 4 | 3 | 7
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race and Ethnicity: African American or Black | 12 | 10 | 22
  Race and Ethnicity: American Indian or Alaskan Native | 0 | 1 | 1
  Race and Ethnicity: Hispanic or Latino(a) | 20 | 24 | 44
  Race and Ethnicity: Multiracial | 2 | 0 | 2
  Race and Ethnicity: White | 1 | 0 | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 35 | 35 | 70

OUTCOME MEASURES:

1. Primary Outcome: Hedonic Liking of Study Foods
Description: Liking of study foods will be measured by showing the name and picture of the meal or ingredient bundle and asking participants to respond to a hedonic 9-point bipolar scale (this scale does not have an official name or title, therefore, 9-point hedonic liking scale can be considered the unabbreviated scale name). The scale has four measures of liking (6-9) and four measures of dislike (1-4) and a neutral "neither like nor dislike" (5). A higher score = more liking of the food. The average of all hedonic liking ratings for each meal was taken to create a hedonic liking score across meals.
Time Frame: 14-days
Population: There were anonymous qualitative interviews conducted with food pantry staff as a separate aim of this study. Food Pantry staff enrolled are not part of the pilot randomized controlled trial (RCT) for which this outcome measure is analyzed since out of the total participants enrolled, only the pantry clients are part of the RCT and the pantry clients who completed this study were analyzed for this outcome. So Food Pantry staff is not included as a separate arm here for this outcome.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | No Prep Ready-to-eat Meals | Ingredient Bundles (e.g. Meal Kits)
Number analyzed (Participants) | 31 | 35
score on a scale | 7.2 (0.9) | 7.2 (1.1)

2. Primary Outcome: Satisfaction of Study Foods
Description: Satisfaction items were adapted from previously validated food pantry client satisfaction surveys (e.g., "How satisfied are you with the amount/variety/frequency of food that you and others in your household receive at this food pantry?") (Dunmire M. Level of satisfaction among food pantry clients, staff/volunteers, and directors and its association with client choice in food pantry layouts. South Dakota State University; 2019.). Response options were "Strongly agree" "Agree" "Disagree" and "Strongly disagree". The items were summed to create an Intervention Satisfaction variable with the lowest possible score of 4 if all responses were "Strongly disagree" and the highest possible score of 20 if all responses were "Strongly agree."
Time Frame: 14-days
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | No Prep Ready-to-eat Meals | Ingredient Bundles (e.g. Meal Kits)
Number analyzed (Participants) | 31 | 35
score on a scale | 15.74 (2.70) | 17.29 (2.31)

3. Secondary Outcome: Perceived Diet Quality
Description: Perceived dietary quality will be measured using a single validated item that asks participants to rate their overall diet quality as "excellent," "very good," "good," "fair," or "poor" (5 = Excellent, 1 = Poor). Perceived diet quality is the scale title.
Time Frame: 14-days
Population: as for outcome 1
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | No Prep Ready-to-eat Meals | Ingredient Bundles (e.g. Meal Kits)
Number analyzed (Participants) | 31 | 35
units on a scale | 3.10 (.18) | 3.4 (.16)

4. Other Pre Specified Outcome: Fruit and Vegetable Frequency
Description: Fruit & Vegetable Screener from the Eating at America's Table Study (EATS) - this is the measure title. Information on how to score the measure can be found at cancer.gov (https://epi.grants.cancer.gov/diet/screeners/fruitveg/instrument.html). The measure is cups of fruits and vegetables per day. A higher number is better.
Time Frame: 14-days
Population: as for outcome 1
Measure: Mean (Standard Error); unit: cups of fruits and veg per day
Arm/Group | No Prep Ready-to-eat Meals | Ingredient Bundles (e.g. Meal Kits)
Number analyzed (Participants) | 31 | 35
cups of fruits and veg per day | 2.81 (2.45) | 3.17 (2.11)

ADVERSE EVENTS:
Time Frame: Adverse event data were collected over 1 month - the duration of participation (two weeks) and two weeks following. However, no adverse events were anticipated or reported.
Description: Pantry staff Group (15 count) is not included in the Adverse Event (AE) Table since they were not monitored for AEs and no AE data were not collected from them. They were not assessed for adverse events. They completed anonymous interviews only. They were not randomized. They did not receive an intervention.
Arm/Group | No Prep Ready-to-eat Meals | Ingredient Bundles (e.g. Meal Kits)
All-Cause Mortality (participants affected / at risk) | 0/35 | 0/35
Serious Adverse Events (participants affected / at risk) | 0/35 | 0/35
Other Adverse Events (participants affected / at risk) | 0/35 | 0/35

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-08-30): https://cdn.clinicaltrials.gov/large-docs/10/NCT05593510/Prot_SAP_000.pdf
  • Informed Consent Form (2023-02-02): https://cdn.clinicaltrials.gov/large-docs/10/NCT05593510/ICF_001.pdf